CLINICAL TRIAL: NCT01327976
Title: A Randomized, Double Blind Sham Controlled Clinical Trial to Evaluate the Safety and Efficacy of vBloc Therapy Delivered by the Maestro Rechargeable System for the Treatment of Obesity
Brief Title: The Safety and Efficacy of vBloc Therapy Delivered by the Maestro Rechargeable System for the Treatment of Obesity
Acronym: ReCharge
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ReShape Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDE G070025
Record Dates: First submitted 2011-03-31; First posted 2011-04-04 (Estimated); Results first posted 2016-05-27 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Obesity
Keywords: Obesity; Bariatric surgery; Excess weight loss; Vagus nerve; Vagal blocking; vBloc Therapy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vBloc (Active Device) (Active Comparator): The treatment group will receive a functional device that will deliver charge to the vagus nerve during the study period
  Interventions: Device: vBloc (Active Device)
- Sham (Non-active Device) (Sham Comparator): The control group will receive a functional, but non-active device that will deliver no charge to the vagus nerve during the study period
  Interventions: Device: Sham (Non-active Device)

INTERVENTIONS:
Device: vBloc (Active Device) — Active device will deliver vBloc Therapy
  Other Names: Maestro® Rechargeable System
  Arms: vBloc (Active Device)
Device: Sham (Non-active Device) — Functional non-active control device will deliver no vBloc Therapy
  Other Names: Maestro® Rechargeable System
  Arms: Sham (Non-active Device)

SUMMARY:
The study evaluated the safety and efficacy of the vBloc Therapy delivered by the Maestro Rechargeable System compared to a sham control for the treatment obesity. The Maestro Rechargeable System delivers intermittent, electrical blocking signals to the anterior and posterior trunks of the intra-abdominal vagus nerve (termed vBloc Therapy) and is designed to reduce sensations of hunger and produce satiety leading to weight loss. After approval from the institutional review board, subjects provided written consent and were randomized in a 2 to 1 allocation to vBloc group (with laparoscopic placement of the leads and neuroregulator) or the sham group (placement of a custom sham neuroregulator only) on double-blinded basis. Both groups received similar diet and exercise counseling. Weight, adverse events, clinical laboratories, ECGs, eating questionnaires and quality of life data were evaluated throughout the 12 month study duration.

DETAILED DESCRIPTION:
The Maestro® Rechargeable System is a neuromodulation system.

All subjects will be randomized in a 2:1 allocation to vBloc or Sham.

All subjects will be followed through the 12-month follow-up visit. Subjects in the Sham group who choose to have an active device will undergo a second surgery to receive the active device after study unblinding.

ELIGIBILITY:
Inclusion criteria

1. Signed informed consent
2. Body mass index (BMI) ≥ 40 kg/m2 to 45 kg/m2 or BMI ≥ 35 kg/m2 to 39.9 kg/m2 with one or more obesity related co-morbid conditions. Co-morbid conditions may include one or more of the following:

   * Type 2 diabetes mellitus as defined in inclusion criteria #5 (limited to 10% of randomized subjects)
   * Hypertension as defined by systolic pressure ≥140 mmHg and/or diastolic pressure ≥90 mmHg a) treated or untreated with systolic ≥140 mmHg or diastolic ≥90 mmHg or b) treated with systolic <140 mmHg and diastolic <90 mmHg
   * Dyslipidemia as defined by total cholesterol ≥200 or LDL ≥130 a) treated or untreated with total cholesterol ≥200 or LDL ≥130 or b) treated with total cholesterol <200 or LDL <130
   * Sleep apnea syndrome (confirmed by overnight p02 studies)
   * Obesity-related cardiomyopathy
3. Females or males Note: females of child-bearing potential must have a negative urine pregnancy test at Screen and also within 14 days of implant procedure followed by physician-approved contraceptive regimen for the duration of the study period.
4. 18-65 years of age inclusive.
5. Type 2 diabetes mellitus subjects:

   * Glycosylated hemoglobin (HbA1c) 7.0 - 10.0 % inclusive at screening visit. (Undiagnosed subjects that are found to have a HbA1c value between 7-10% at screening must see their primary physician for diagnosis and medical treatment before continuing in trial)
   * Onset: 12 years or less since initial diagnosis.
   * Currently not using insulin therapy, GLP-1 (glucagon-like peptide-1) receptor agonists (e.g., exenatide, liraglutide) for diabetes treatment and have not been on these treatments in the past 6 months.
   * Creatinine within normal reference range.
   * No history of proliferative retinopathy.
   * No history of peripheral neuropathy.
   * No history of autonomic neuropathy.
   * No history of coronary artery disease, with or without angina pectoris.
   * No history of peripheral vascular disease.
6. Failure to respond to supervised diet/exercise program(s) in which the subject was engaged within the last five years.
7. Ability to complete all study visits and procedures.

Exclusion criteria

1. Concurrent chronic pancreatic disease.
2. History of Crohn's disease and/or ulcerative colitis.
3. History of bariatric surgery, fundoplication, gastric resection or major upper-abdominal surgery (acceptable surgeries include cholecystectomy, hysterectomy).
4. History of pulmonary embolism or blood coagulation disorders.
5. Clinically significant hiatal hernias (> 5 cm) known from subject's medical record or determined by barium swallow (upper GI x-ray) or upper endoscopy per PI discretion prior to implant.
6. Current cirrhosis, portal hypertension and/or esophageal varices.
7. Intra-operative exclusion: hiatal hernia requiring surgical repair or extensive dissection at esophagogastric junction at time of surgery.
8. Treatment with prescription weight-loss drug therapy within the prior three months and the use of prescription drug therapy or the use of over-the-counter weight loss preparations for the duration of the trial.
9. Smoking cessation within the prior six months.
10. Known genetic cause of obesity (e.g., Prader-Willi Syndrome).
11. Weight loss of more than 10% of body weight in the previous 12 months.
12. Physician-prescribed diet with intent to lose weight prior to surgery (note:

    study subject may continue any personal eating plan they were on prior to study enrollment [see exclusion criterion #24]
13. Current type 1 diabetes mellitus (DM).
14. Current or recent history (within 12 months) of ongoing bulimia.
15. Current alterations in treatment for thyroid disorders (stable treatment regimen for prior three months acceptable).
16. Current alterations in treatment for epilepsy (stable treatment regimen for prior six months acceptable).
17. Current treatment for peptic ulcer disease (previous history acceptable).
18. Chronic (more than 4 weeks of daily use) treatment with narcotic analgesic drug regimens (treatment with non-steroidal anti-inflammatory drugs acceptable).
19. Current alterations in treatment regimens of anti-cholinergic drugs, including tricyclic antidepressants (stable treatment regimen for prior six months acceptable).
20. Current medical condition that, in the opinion of the investigator, would make subject unfit for surgery under general anesthesia or that would be exacerbated by intentional weight loss. Some examples include diagnosis of cancer, recent heart attack, recent stroke, or recent serious trauma.
21. Presence of permanently implanted electrical powered medical device or implanted gastrointestinal device or prosthesis (e.g., pacemakers, implanted defibrillators, neurostimulators etc.).
22. Planned or contemplated use of Magnetic Resonance Imaging (MRI) or oncologic radiation during the course of the trial.
23. Psychiatric disorders (including untreated severe depression, schizophrenia, substance abuse, bulimia nervosa, etc.) or limited intellectual functioning which would potentially compromise the participant's ability to fully comprehend and/or cooperate with the study protocol. Psychiatric disorders will be established by a review of subject's medical history. For depression, a BDI (Beck Depression Inventory) score ≥ 29 will be considered to indicate severe depression.
24. Current, active member of an organized weight loss program (e.g., Weight Watchers, TOPS).
25. Current participant in another weight loss study or other clinical trials.
26. Have a friend or family member who is currently participating or is planning to participate in this clinical trial.
27. Patient reported:

    * inability to walk for about 10 minutes without stopping,
    * feeling of pain in chest when doing physical activity,
    * feeling of pain in chest when not doing physical activity. Note: unless pain in chest in known to be related to upper gastrointestinal disorders such as gastroesophageal reflux disease or heartburn.
28. Clinically significant cardiac rhythm disorder that requires either medical and/or surgical intervention (e.g., paroxysmal or chronic atrial fibrillation).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2011-05; Primary Completion 2013-02 (Actual); Study Completion 2021-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sarr, M.D., Principal Investigator — Mayo Clinic; Charles Billington, M.D., Principal Investigator — University of Minnesota
Locations (10):
- United States (8):
  - HonorHealth (formerly Scottsdale Healthcare Bariatric Center), Scottsdale, Arizona
  - Scripps Clinic Nutrition & Metabolic Research Center, La Jolla, California
  - Stanford University, Stanford, California
  - Tufts Medical Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Oregon Health & Science University, Portland, Oregon
  - Virginia Commonwealth University, Richmond, Virginia
- Australia (2):
  - Institute of Weight Control, Baulkham Hills, New South Wales
  - Adelaide Bariatric Centre, Bedford Park, SA

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Apovian CM, Shah SN, Wolfe BM, Ikramuddin S, Miller CJ, Tweden KS, Billington CJ, Shikora SA. Two-Year Outcomes of Vagal Nerve Blocking (vBloc) for the Treatment of Obesity in the ReCharge Trial. Obes Surg. 2017 Jan;27(1):169-176. doi: 10.1007/s11695-016-2325-7. PMID 27506803
- [Derived] Ikramuddin S, Blackstone RP, Brancatisano A, Toouli J, Shah SN, Wolfe BM, Fujioka K, Maher JW, Swain J, Que FG, Morton JM, Leslie DB, Brancatisano R, Kow L, O'Rourke RW, Deveney C, Takata M, Miller CJ, Knudson MB, Tweden KS, Shikora SA, Sarr MG, Billington CJ. Effect of reversible intermittent intra-abdominal vagal nerve blockade on morbid obesity: the ReCharge randomized clinical trial. JAMA. 2014 Sep 3;312(9):915-22. doi: 10.1001/jama.2014.10540. PMID 25182100

RESULTS

PARTICIPANT FLOW:
Groups:
- vBloc (Active Device): The treatment group will receive a functional device that will deliver charge to the vagus nerve during the study period.
  Active, implantable, intra abdominal vagal blocking medical device (Maestro® Rechargeable System): Active device will deliver vBloc Therapy.
- Sham (Non-active Device): The control group will receive a functional, but non-active device that will deliver no charge to the vagus nerve during the study period.
  Active, implantable, intra abdominal vagal blocking medical device (Maestro® Rechargeable System): Control device will deliver no vBloc Therapy.
Period: Overall Study
Arm/Group | vBloc (Active Device) | Sham (Non-active Device)
Started | 162 | 77
Completed | 154 | 70
Not Completed | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- vBloc (Active Device): The vBloc group will receive a functional device that will deliver charge to the vagus nerve during the study period.
  Active, implantable, intra abdominal vagal blocking medical device (Maestro® Rechargeable System): Active device will deliver vBloc Therapy.
- Sham (Non-active Device): The Sham group will receive a functional, but non-active device that will deliver no charge to the vagus nerve during the study period.
  Active, implantable, intra abdominal vagal blocking medical device (Maestro® Rechargeable System): Control device will deliver no vBloc Therapy.
- Total: Total of all reporting groups
Arm/Group | vBloc (Active Device) | Sham (Non-active Device) | Total
Number analyzed (Participants) | 162 | 77 | 239
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 162 | 77 | 239
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (10) | 47 (9) | 47 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 62 | 203
  Male | 21 | 15 | 36
Region of Enrollment [Number; unit: participants]
  United States | 122 | 60 | 182
  Australia | 40 | 17 | 57

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Experiencing Implant/Revision Procedure, Device or Therapy Related Serious Adverse Events (SAEs).
Description: To demonstrate that the implant/revision procedure, device and therapy related serious adverse event rate in the vBloc group at 12 months post-implant is significantly lower than 15%.
Time Frame: 12 months
Population: An intent-to-treat analysis was performed in the vBloc group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- vBloc (Active Device): The vBloc group received an active, implantable, vagal blocking medical device (Maestro® Rechargeable System) that delivered charge to the intra-abdominal anterior and posterior vagal trunks during the study period
- Sham (Non-active Device): The Sham group received a device that dissipated charges into an electronic circuit within the device with no lead placement. Therefore, no charge was delivered to the vagus nerve during the study period.
Arm/Group | vBloc (Active Device) | Sham (Non-active Device)
Number analyzed (Participants) | 162 | 77
percentage of participants | 3.7 [1.4 to 7.9] | 0 [0 to 0]

2. Primary Outcome: Percentage of Excess Weight Loss (EWL) by Body Mass Index (BMI) Method.
Description: Observe at least a 10% greater excess body weight loss (EWL) from randomization with the Maestro System after 12 months of vBloc Therapy compared to Sham by body mass index (BMI) method. (Body mass index is calculated by dividing body weight (kg) by body height (m) squared (BMI=kg/m2)).
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: percentage of excess weight loss
Groups:
- vBloc (Active Device): The vBloc group will receive a functional device that will deliver charge to the vagus nerve during the study period
  Active, implantable, intra abdominal vagal blocking medical device (Maestro® Rechargeable System): Active device will deliver vBloc Therapy
- Sham (Non-active Device): The Sham group will receive a functional, but non-active device that will deliver no charge to the vagus nerve during the study period
  Active, implantable, intra abdominal vagal blocking medical device (Maestro® Rechargeable System): Control device will deliver no vBlocTherapy
Arm/Group | vBloc (Active Device) | Sham (Non-active Device)
Number analyzed (Participants) | 162 | 77
percentage of excess weight loss | 24.4 [20.8 to 28.1] | 15.9 [11.9 to 19.9]

3. Primary Outcome: Percentage Responder Rate in the Treatment Arm.
Description: The second co-primary effectiveness endpoint was based on responder rates with the following two requirements: (i) at least 55% of vBloc subjects would achieve a %EWL of at least 20%; and (ii) at least 45% of vBloc subjects would achieve a %EWL of at least 25%.
Time Frame: 12 months
Measure: Number; unit: percentage of subjects
Arm/Group | vBloc (Active Device) | Sham (Non-active Device)
Number analyzed (Participants) | 162 | 77
percentage of subjects
  % of subjects achieving an EWL of at least 20% | 52.5 | 32.5
  % of subjects achieving an EWL of at least 25% | 38.3 | 23.4

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- vBloc (Active Device): The treatment group will receive a functional device that will deliver charge to the vagus nerve during the study period.
  Active, implantable, intra abdominal vagal blocking medical device (Maestro® Rechargeable System): Active device will deliver vBlocTherapy.
Arm/Group | vBloc (Active Device) | Sham (Non-active Device)
Serious Adverse Events (participants affected / at risk) | 26/162 | 4/77
Other Adverse Events (participants affected / at risk) | 128/162 | 53/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | vBloc (Active Device) (N=162) | Sham (Non-active Device) (N=77)
Neuroregulator malfunction (Surgical and medical procedures) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gallbladder disease (Hepatobiliary disorders) | 2 (2) | 0 (0)
Emesis/vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain, neuroregulator site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 0 (0)
Cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) — Subject not implanted
Generalized ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-operative oozing (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Allergic reaction (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infection, other (Infections and infestations) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain, abdominal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain, other (General disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Worsening back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | vBloc (Active Device) (N=162) | Sham (Non-active Device) (N=77)
Pain, neuroregulator site (Skin and subcutaneous tissue disorders) | 65 (78) | 32 (37)
Other (General disorders) | 90 (157) | 40 (62)
Heartburn/dyspepsia (Gastrointestinal disorders) | 42 (46) | 4 (4)
Pain, other (General disorders) | 80 (136) | 28 (36)
Pain, abdominal (Gastrointestinal disorders) | 25 (32) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 14 (14) | 1 (1)
Eructation/belching (Gastrointestinal disorders) | 13 (13) | 0 (0)
Incision pain (Surgical and medical procedures) | 12 (13) | 7 (7)
Chest pain (General disorders) | 10 (10) | 3 (4)
Wound redness or irritation (Skin and subcutaneous tissue disorders) | 7 (7) | 5 (5)
Cold/flu/respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 70 (121) | 33 (58)
Constipation (Gastrointestinal disorders) | 24 (24) | 13 (15)
Headache (General disorders) | 21 (24) | 8 (9)
Out of range lab values (Metabolism and nutrition disorders) | 20 (23) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 18 (19) | 4 (4)
Trauma (General disorders) | 15 (19) | 11 (18)
Infection, other (Infections and infestations) | 15 (18) | 11 (12)
Nausea (Gastrointestinal disorders) | 13 (15) | 3 (3)
Emesis/vomiting (Gastrointestinal disorders) | 11 (12) | 6 (6)
Reaction to medicines (General disorders) | 10 (12) | 6 (6)
Anxiety (Psychiatric disorders) | 11 (11) | 3 (3)
Dizziness (General disorders) | 10 (10) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days